CLINICAL TRIAL: NCT05751967
Title: A Prospective, Multi-center, Randomized, Double-blind, Placebo-controlled Study: Fenofibrate Combined With Ursodeoxycholic Acid in Subjects With Primary Biliary Cholangitis and an Inadequate Response to Ursodeoxycholic Acid
Brief Title: Fenofibrate Combined With Ursodeoxycholic Acid in Subjects With Primary Biliary Cholangitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20222274-C-1
Record Dates: First submitted 2022-12-13; First posted 2023-03-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 1 tablet/ day
  Interventions: Drug: Placebo Combined With Ursodeoxycholic Acid
- Fenofibrate (Experimental): 200 mg/day
  Interventions: Drug: Fenofibrate Combined With Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Placebo Combined With Ursodeoxycholic Acid — 1 tablet/ day
  Other Names: UDCA 13-15mg/kg/d
  Arms: Placebo
Drug: Fenofibrate Combined With Ursodeoxycholic Acid — 200 mg/day
  Other Names: UDCA 13-15mg/kg/d
  Arms: Fenofibrate

SUMMARY:
Current treatment guidelines recommend ursodeoxycholic acid (UDCA) as the first-line treatment for new-diagnosed primary biliary cholangitis (PBC) patients. However, up to 40% patients are insensitive to UDCA monotherapy, and evaluation of UDCA response at 12 months may result in long period of ineffective treatment. We aimed to develop a new criterion to reliably identify non-response patients much earlier. Recently, our team designed and validated a new early criterion for distinguishing high-risk PBC patients in a Chinese population for the first time. Our data indicated that PBC patients with ALP ≤ 2.5 × ULN, AST ≤ 2 × ULN, and TBIL ≤ 1 × ULN (Xi'an criterion) after 1 month UDCA treatment were likely to have better prognosis. It can be readily applied in the rapid identification of PBC patients who require additional therapeutic approaches. However, whether it is reasonable to apply it to the response definition of clinical research, and the guidance of PBC management and choice of second-line treatment, further research is needed.

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled, parallel-group study that will assess the efficacy and safety of fenofibrate in patients with PBC who had an inadequate biochemical response to UDCA, as defined by the Xi'an criteria. Fenofibrate or placebo 200 mg will be daily administered in combination with UDCA 13-15 mg/kg/d for 48 months. Patient safety will be monitored. Primary end-point will be the percentage of patients with a complete normalization of the ALP and TBIL. Secondary endpoints will include the percentage of drug-related adverse events, survival rates without liver transplantation or liver decompensation, time course of non-invasive liver fibrosis measurements (LSM), time course of endoscopic, ultrasound, and biochemical features of portal hypertension, time course of pruritus and of quality of life using validated scales.

ELIGIBILITY:
Inclusion Criteria:

* Must have provided written informed consent;
* Age 18-75 years;
* BMI 17-28 kg/m2
* Male or female with a diagnosis of PBC, by at least two of the following criteria:

  * History of AP above ULN for at least six months;
  * Positive AMA titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies;
  * Documented liver biopsy result consistent with PBC.
* Incomplete response to UDCA defined by Xi'an criteria (ALP >2.5× ULN, AST>2×ULN or TBIL>1×ULN) after UDCA treatment for 4-6 weeks with at least one abnormal test in ALP or TBIL.

Exclusion Criteria:

* History or presence of other concomitant liver diseases.
* ALT/AST > 5×ULN, TBIL > 3×ULN.
* If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
* Allergic to fenofibrate or ursodeoxycholic acid.
* Taking hepatotoxic drugs (e.g., dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) for more than 2 weeks within 6 months, and long-term hormonal users.
* Recurrent variceal bleeding, poorly controlled hepatic encephalopathy or refractory ascites.
* Patients with a history of severe cardiac, cerebrovascular, renal, respiratory disease or functional failure, and psychiatric disorders (including those due to alcohol and drug abuse).
* Creatinine >1.5×ULN and creatinine clearance <60 ml/min.
* Currently using statins (such as pravastatin, fluvastatin, and simvastatin), other fibrates (such as gemfibrozil and bezafibrate), and drugs structurally similar to fenofibrate (like ketoprofen).
* Planned to receive an organ transplant or an organ transplant recipient.
* Needing Liver transplantation within 1 year according to the Mayo Rick score.
* Any other condition(s) that would compromise the safety of the subject or compromise the quality of the clinical study, as judged by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete biochemical response | 48 weeks
  The normalisation of Alkaline Phosphatase (ALP) and total bilirubin (TBIL).

SECONDARY OUTCOMES:
Percentage of patients having complete biochemical response | 4, 12, 24, 36, and 48 weeks
  The normalisation of Alkaline Phosphatase (ALP) and total bilirubin (TBIL) at 4, 12, 24, and 36 weeks.
Assessment of the fatigue and the quality of life | 4, 12, 24, 36, and 48 weeks
  Change from baseline in primary biliary cholangitis -40 (PBC-40) quality of life (QoL) questionnaire scores.
Assessment of the fatigue and the quality of life | 4, 12, 24, 36, and 48 weeks
  Change from baseline in pruritus as assessed by Visual Analogue Scale (VAS) total score for fatigue and pruritus.
Evolution of the biological markers of the hepatic function or being in the usual prognostic scores | 4, 12, 24, 36, and 48 weeks
  Mayo score at 4, 12, 24, 36, and 48 weeks
Evolution of the biological markers of the hepatic function or being in the usual prognostic scores | 4, 12, 24, 36, and 48 weeks
  Child-Puch score at 4, 12, 24, 36, and 48 weeks
Evolution of the biological markers of the hepatic function or being in the usual prognostic scores | 4, 12, 24, 36, and 48 weeks
  MELD score at 4, 12, 24, 36, and 48 weeks
Evolution of the biological markers of the hepatic function or being in the usual prognostic scores | 48 weeks
  GLOBE-PBC score at 48 weeks
Evolution of the biological markers of the hepatic function or being in the usual prognostic scores | 48 weeks
  UK-PBC score at 48 weeks
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of creatinine
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of Blood urea nitrogen
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of creatine kinase
Percentage of patients having biological or clinical adverse events | 4, 12, 24, 36, and 48 weeks
  Increase of ALT and AST.
Survival without transplantation and hepatic impairment | 48 weeks
  Occurrence of ascites, variceal bleeding, hepatic encephalopathy, liver-transplantation, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, Doctor, Principal Investigator — The First Affiliated Hospital of Air Force Medicial University
Locations (7):
- China (7):
  - The second hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Ying han, Xi'an, Shaanxi
  - Sichuan Provincial People's Hospital,, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No